CLINICAL TRIAL: NCT03762811
Title: Post-Market Clinical Investigation of NanoFUSE® Bioactive Matrix
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NanoFUSE Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR-00002
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Bone; Degeneration
Keywords: Demineralized Bone Matrix; Bone Graft; Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- NanoFUSE® PMCF (Other): NanoFUSE® Bioactive Matrix will be implanted according to labeling and the intended surgical treatment plan of the surgeon.
  Interventions: Device: NanoFUSE® Bioactive Matrix

INTERVENTIONS:
Device: NanoFUSE® Bioactive Matrix — NanoFUSE® is placed into bony voids or gaps of the skeletal system that are not intrinsic to the stability of the bony structure.

SUMMARY:
This purpose of this study is to determine fusion rates and compare clinical outcomes of the NanoFUSE® Bioactive Matrix during post-market clinical use.

DETAILED DESCRIPTION:
NanoFUSE® is indicated to be placed into bony voids or gaps of the skeletal system that are not intrinsic to the stability of the bony structure (i.e. the posterolateral spine and pelvis). These defects may be surgically created osseous defects or osseous defects created from traumatic injury to bone. NanoFUSE® must be used with autograft as a bone graft extender in the posterolateral spine and pelvis. This product provides a bone graft substitute that remodels into the recipient's skeletal system.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature
* Medically suitable for surgical management and the use of NanoFUSE® Bioactive Matrix consistent with product labeling
* Psychosocially, mentally, and physically able to fully comply with the protocol, including the post-operative regimen, requires follow-up visits, filling out required forms, and the ability to understand and give written informed consent
* Retrospective data collection must be allowed by the IRB and all information deidentified

Exclusion Criteria:

* Previous fusion surgery of the proposed site
* Use of chronic medications known to affect the skeleton (e.g. glucocorticoid usage > 10mg/day)
* Pregnant or female intending to become pregnant during this study period
* Obesity (BMI >40kg/m2)
* Systemic infection or infection at the surgical site
* Current or past substance abuse
* Poor general healthy or any concurrent disease process that would place the patient in excessive risk to surgery (e.g. significant circulatory or pulmonary problems, cardiac disease
* Medical condition that would interfere with post-operative assessments and care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Radiographic Success that indicates patient achieving fused or probably fused status. | 12 months
  at 12 months

SECONDARY OUTCOMES:
Overall patient success | 12 months postoperatively
  Overall patient success will be based on all clinical and radiographic evaluation